CLINICAL TRIAL: NCT07107763
Title: Investigation of the Effects of Short Foot Exercise and Mobilization in Young Adults With Pes Planus
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Kirsehir Ahi Evran Universitesi (Other)
Responsible Party: Principal Investigator, Muhammed Samed DALAKÇI, Principal Investigator, Kirsehir Ahi Evran Universitesi
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: MSDLKCİ
Record Dates: First submitted 2025-07-19; First posted 2025-08-06 (Actual); Last update posted 2025-12-18 (Actual); Status verified 2025-12

CONDITIONS: Pes Planus
MeSH Terms: conditions — Flatfoot

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Short foot exercise (Active Comparator): A program consisting of short foot exercises will be implemented for the short foot exercise group, with three sessions per week over a period of six weeks. Each session will begin with stretching exercises, followed by the short foot exercises.
  Interventions: Other: Mobilization
- Mobilization (Active Comparator): The mobilization group will undergo a program consisting of 3 sessions per week for a duration of 6 weeks. The sessions will begin with stretching exercises, followed by subtalar joint mobilization.
  Interventions: Other: short foot exercise
- short foot exercise and mobilization (Experimental): The combined intervention used in this group will include both of the approaches applied in the other two groups.
  Interventions: Combination Product: Short foot exercise and mobilization

INTERVENTIONS:
Other: short foot exercise — The short foot exercise group will receive stretching exercises and short foot exercises, administered three sessions per week for a duration of six weeks.
  Arms: Mobilization
Other: Mobilization — The mobilization group will undergo a program consisting of 3 sessions per week for a duration of 6 weeks. The sessions will begin with stretching exercises, followed by subtalar joint mobilization.
  Arms: Short foot exercise
Combination Product: Short foot exercise and mobilization — The combined intervention used in this group will include both of the approaches applied in the other two groups.
  Arms: short foot exercise and mobilization

SUMMARY:
Pes Planus (PP) is a foot deformity characterized by a lower-than-normal medial longitudinal arch. Individuals diagnosed with PP experience various challenges in daily life. Among these challenges are limitations in balance and movement skills. To reduce the effects of PP, several treatment approaches are preferred. These interventions are generally categorized into surgical and conventional treatments. Among conservative approaches, the short foot exercise is one of the most fundamental and commonly used methods. This exercise aims to strengthen the intrinsic muscles of the foot to support the arch. In addition to the short foot exercise, other exercises such as towel scrunching and toe spreading are also used in the management of PP. However, when looking at the treatment options for PP, studies examining the use and effects of joint mobilization are limited. The present study aims to investigate the effects of subtalar joint mobilization, short foot exercises, and the combined application of these interventions in individuals with PP. This approach is based on findings that subtalar joint mobilization has positive effects on balance in individuals with balance impairments.

ELIGIBILITY:
Inclusion Criteria:

* To be diagnosed with flexible pes planus

Exclusion Criteria:

* Having other comorbidities

Ages: 18 Years to 30 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 45 (Actual)
Dates: Start 2025-09-26 (Actual); Primary Completion 2025-12-17 (Actual); Study Completion 2025-12-17 (Actual)

PRIMARY OUTCOMES:
Vertical Jump Test | From enrollment to the end of treatment at 6 weeks
Shuttle Run Test | From enrollment to the end of treatment at 6 weeks

SECONDARY OUTCOMES:
Standing Broad Jump Test | From enrollment to the end of treatment at 6 weeks
Biodex Balance Assessment | From enrollment to the end of treatment at 6 weeks

CONTACTS AND LOCATIONS:
Locations (1):
- Kırşehir Ahi Evran University, Kırşehir, Turkey (Türkiye)